CLINICAL TRIAL: NCT04604340
Title: Radial Versus Femoral Arterial Access for Cerebral Angiography in Adolescents: A Randomized-controlled Study
Brief Title: Radial Versus Femoral Arterial Access for Cerebral Angiography in Adolescents
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: insufficient enrolment-radial access for neuroangiography is now accepted as clinical standard.
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Prakash Muthusami, Neurointerventionist, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1000065604
Record Dates: First submitted 2020-10-01; First posted 2020-10-27 (Actual); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Procedural Related Injuries and Complications Nec; Patient Satisfaction
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- transfemoral access (Active Comparator): control
  Interventions: Procedure: transradial access for neuroangiography; Procedure: transfemoral access for neuroangiography
- transradial access (Active Comparator): case
  Interventions: Procedure: transradial access for neuroangiography; Procedure: transfemoral access for neuroangiography

INTERVENTIONS:
Procedure: transradial access for neuroangiography — The choice of right vs left radial artery approach would be determined by the vessels that require the highest quality of imaging (e.g. if the left vertebral artery is key to diagnosis, a left radial approach would be chosen, otherwise a right radial approach would be likely most appropriate) - this decision is at the discretion of the interventionist.
Procedure: transfemoral access for neuroangiography — By convention, femoral access will be obtained on the right side, unless there is overlying disease or vessel abnormality detected by ultrasound/Doppler, as is usual clinical practice.

SUMMARY:
This study will compare radial vs femoral access for angiography in adolescents. Neuroangiography and neurointerventions are predominantly performed via femoral access, which has several limitations and complications - pain and discomfort, arterial occlusion, retroperitoneal hemorrhage, activity limitations, and increased admissions. Transradial angiography has shown promise to circumvent these problems, but this has not been studied in children, whose unique anatomical and physiological aspects require that this be evaluated rigorously.

DETAILED DESCRIPTION:
Specific Aims:

Angiography in interventional radiology is still most commonly performed through femoral arterial access, wherein patients are committed to invasive procedures through access at their groin, which entails anxiety, embarrassment, pain and discomfort, the inability to resume normal activities for a week, serious complications like retroperitoneal hemorrhage, and increased hospital admissions. Angiography through access at the wrist (transradial angiography) has been shown with some recent data to circumvent these complications and, in general, provide a more satisfactory and safe patient experience. Although transradial angiography has been rapidly accepted by some operators, especially in Cardiology, the absence of evidence for technical details and safety has resulted in much debate in the literature and in recent conferences. Specifically, there is no literature reported in children. The benefits of a method which would allow mobility immediately after the procedure in children are self-evident - this would potentially result in less rebleeds, require little or no sedation, allow sitting up and feeding, and allow parents to interact with their child and feel more comfortable. On the flip side, the feasibility and potential complications in children are unknown, and thus this technique cannot be integrated into clinical practice without interrogating this. This should be ideally performed in a high volume pediatric center with expertise in not only pediatric neuroangiography, but also for minimally invasive arterial access with interventional radiology, to minimize complications. Given the size consideration of arteries in children, we believe a good start point for this study would be with adolescent children.

The Investigator's objective is to provide the highest level of evidence (RCT data) for feasibility, safety and technique of transradial angiography in adolescents, by comparing it against the current gold standard, trans-femoral angiography. This will provide data for subsequent practice guidelines.

This study will be performed in a tertiary pediatric institution, with collaboration between interventional radiologists, neuroradiologists, pediatricians, neurosurgeons, technologists, statisticians, research co-ordinators and imaging physicists. A large number of clinical cases, established pipelines for clinical workflow and research collaborations and imaging laboratories with personnel and students would enable us to successfully complete this project in a timely manner.

Neuroangiography and neurointerventions are predominantly performed via femoral access, which has several limitations and complications - pain and discomfort, arterial occlusion, retroperitoneal hemorrhage, activity limitations, and increased admissions. Transradial angiography has shown promise to circumvent these problems, but this has not been studied in children, whose unique anatomical and physiological aspects require that this be evaluated rigorously.

Primary aim:

To evaluate procedural comfort and acceptance of transradial vs. transfemoral neuroangiography in a cohort of randomized adolescent children. This will be performed using patient self-reported pain and satisfaction scores.

Secondary aim:

1. To evaluate procedural safety for transradial vs. transfemoral neuroangiography in a cohort of adolescent children. This will be performed by comparing fluoroscopy time and dose, procedural and long-term complication rates, study completeness and admission times.

Methods: Children (8-18 years) scheduled for supra-aortic angiography will be approached to participate. Inclusion cut-offs: radial artery ultrasound diameter >20mm and positive Allen test. For 95% power (primary aim), the Investigator will require a sample size of 56. Neuroangiography will be performed as clinically indicated, with collection of demographics, procedural details (screening time, radiation dose, completeness and complications) and post-procedural details (visual analog pain scale, satisfaction score, complications). A Data & Safety Monitoring board will audit the trial.

Outcome Measures: Self-reported scores will be compared between groups for procedural acceptance; complications will be compared for procedural safety.

Significance: 1) This study will provide the highest level evidence regarding role and safety of transradial neuroangiography in children. 2) Subsequent development of practice guideline recommendations for a standardized protocol for transradial angiography in children.

ELIGIBILITY:
Inclusion Criteria:

1. Age 8-18 years
2. Planned cerebral or supra-aortic angiography for clinical reason
3. Positive modified Allen's test using a pulse oximeter on the index finger.
4. Radial artery axial maximal diameter of > 2.0 mm measured on a cross-sectional B-mode ultrasound of the distal radial artery, 2-3 cm proximal to the radial styloid, at the anticipated needle puncture site -

Exclusion Criteria:

1. Age <8 years
2. Radial artery internal maximal of diameter 2.0 mm or less (measured on cross-sectional ultrasound 2-3 cm proximal to the radial styloid at the planned puncture site) - these patients would be converted to femoral access without radial artery puncture but would be assessed in the radial artery group as part of an intention-to-treat analysis.
3. Conversion to intervention (as opposed to diagnostic cerebral angiogram) during the procedure, as this will likely require a larger (femoral) access sheath; again such patients will still be assessed as part of the intention-to-treat analysis.
4. Failed modified Allen's test with pulse oximetry

   -

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2020-09-22 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Procedural access-related complications | intraprocedural
  access-related complications
Procedural access-related complications | 30 days
  access-related complications
Procedural access-related complications | 365 days
  access-related
other Procedural complications | intra procedural
  other procedural complications
other Procedural complications | 30 days
  other procedural complications
other Procedural complications | 365 days
  other procedural complications
Procedural complications-completion rate | intraprocedural
  study completion rate
Procedural complications - long term | 30 days
  long term complications
pain score | 3 hours post-procedure
  visual analog scale VAS with 0=no pain, and 10 being worst pain
patient/parent satisfaction score | 3 days post-procedure
  modified Likert scale-0=unsatisfied, and 5=completely satisfied

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital for Sick Children, Toronto, Ontario, Canada